CLINICAL TRIAL: NCT02818166
Title: Magnetic Resonance Neurological Evaluation After Right Mini-thoracotomy Mitral Valve Surgery: Trans-thoracic Versus Endoaortic Clamp
Brief Title: Magnetic Resonance Imaging for Cerebral Embolization During Minimal Invasive Mitral Valve Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Cristina Barbero, Cardiothoracic Surgeon, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Turin University
Record Dates: First submitted 2016-01-05; First posted 2016-06-29 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Neurological Complications; Mitral Valve Insufficiency
Keywords: magnetic resonance; right mini-thoracotomy
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoaortic Clamp (Experimental): Right mini-thoracotomy mitral valve surgery with retrograde perfusion and endoaortic balloon clamp
  Interventions: Procedure: Mitral valve surgery
- Transthoracic Clamp (Active Comparator): Right mini-thoracotomy mitral valve surgery with retrograde perfusion and transthoracic clamp.
  Interventions: Procedure: Mitral valve surgery

INTERVENTIONS:
Procedure: Mitral valve surgery — Right mini-thoracotomy mitral valve replacement/repair.

SUMMARY:
The purpose of this study is to prospectively evaluate major and minor neurologic events in patients undergoing right mini-thoracotomy mitral valve surgery and to compare different aortic clamping techniques; specifically, the endoaortic balloon with retrograde perfusion (Endoreturn) and the transthoracic clamp with retrograde perfusion. Major neurologic events will be evaluate through standard neurologic evaluation; minor neurologic events will be evaluate through magnetic resonance (MR) assessment.

The first aim of the study is to determine the number and impact of microembolic events during right mini-thoracotomy mitral valve surgery on clinical neurological status and on MR evaluation. The investigators also aim to determine if different techniques of aortic clamping may impact on early outcome.

Study hypothesis: despite recent concerns arising about endoaortic balloon with retrograde perfusion, the investigators expect to show equivalence in term of safety and effectiveness of this technique compared with the transthoracic clamp in a selected population.

DETAILED DESCRIPTION:
The incidence of neurologic events in right mini-thoracotomy mitral valve surgery compared with that of conventional surgery is a controversial issue and has been extensively studied. In the meta-analysis published by Modi et al, equal occurrence of neurologic events between patients who underwent MIMVS and those who underwent a median sternotomy was found. Conversely, the Thoracic Surgeons Adult Cardiac database and the Cleveland Clinic group concluded that the risk of stroke is significantly higher in the less invasive group.

Moreover, recent data have suggested that retrograde arterial perfusion, particularly in patients with severe arch/ascending aortic atherosclerosis, could be the source of the significant increase in the incidence of cerebral complications. The meta-analysis of Cheng, documents a 1.79 fold increase in the risk of stroke in the right thoracotomy group, but on subgroup analysis this appeared driven by a higher stroke risk in those studies reporting endoaortic balloon occlusion and not transthoracic clamping. Murzi et al. report a 4.28 fold increase in stroke risk with RAP in 1280 primary MIMVS patients. Grossi and colleagues show that the only significant risk factor for neurologic event was the use of retrograde perfusion in high-risk patients with aortic disease.

The purpose of this randomized blinded study is to prospectively evaluate major and minor neurologic events in patients undergoing right thoracotomy mitral valve surgery with retrograde perfusion and endoaortic balloon clamp (Endoreturn) or transthoracic clamp. Major neurologic events will be evaluate through standard neurologic evaluation; minor neurologic events will be evaluate through magnetic resonance assessment.

MR evaluation will be performed by blinded radiologists. MR will be performed with a 3T system (Philips INGENIA 3T). The protocol includes conventional sequences for the morphological and quantitative assessment (3D-FLAIR, 3D-T1-TSE, DWI, T2-FFE) and non conventional sequences for the white matter microstructural evaluation (Diffusion Tensor Imaging - DTI with fractional anisotropy and mean diffusivity). No contrast enhanced will be used.

Patients who have no contraindications will undergo cerebral MR before surgery as baseline assessment. Then, they will be randomized in one of the 2 groups.

If no contraindications arise in the postoperative period (eg definitive pacemaker implantation), patients will undergo cerebral MR before the discharge, to highlight the presence of new ischemic lesions, even clinically silent.

After 6 months, patients who developed new ischemic lesions revealed by the post-operative cerebral MR will repeat a new MR to assess evolution of cerebral damage Neurologic assessment will be performed by blinded specialists of the Neurology Department.

Type of the study:

Single center randomized blinded study that will be performed at the University of Turin, Città della Salute e della Scienza Hospital and will include:

Cardiac Surgery department. Neuroradiology department.

Aims of the study:

To determine the incidence of new lesions on pre-discharge MR in patients undergoing right mini-thoracotomy mitral valve surgery according to different aortic clamping techniques.

To assess the correlation between clinical neurological peri-procedural events (TIA, Stroke), and the occurrence of new lesions on pre-discharge MR.

To assess the evolution of new cerebral ischemic lesions between pre-discharge MR and follow-up MR (more than 6 months later).

To the investigators knowledge this is the first randomized blinded study that will compare two right mini-thoracotomy techniques for mitral valve surgery on a selected population (without risk factors for neurological events) with MR.

The result of this study will be able to allow surgeons to choose the best and less dangerous method in case of mini-invasive operations. This could rapresent a fundamental step in confirming the efficacy and safety of mini-invasive approaches for mitral valve surgery and resulting, in addition, in the reduction of the costs of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years.
* Indication for elective mitral valve surgery +/- tricuspid valve surgery through right mini-thoracotomy.
* No contraindication for MR

Exclusion Criteria:

* Neuro-cognitive diseases;
* Peripheral vascular disease;
* Atrial fibrillation;
* PFO o interatrial defect;
* Previous Stroke;
* Autoimmune diseases;
* Neoplastic diseases;
* Migraine;
* Celiac disease;
* Alchool or drug abuse;
* Contraindication for MR.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
MR microembolization | untill 3 days after surgical procedure
  To determine the incidence of new lesions on pre-discharge MR in patients undergoing right mini-thoracotomy mitral valve surgery according to different aortic clamping techniques.
Clinical events and MR outcome correlation | untill 3 days after surgical procedure
  To assess the correlation between clinical neurological peri-procedural events (TIA, Stroke), cognitive / neuropsychological status and the occurrence of new lesions on pre-discharge MR.

SECONDARY OUTCOMES:
Evolution of MR lesions | 3 month follow up
  To assess the evolution of new cerebral ischemic lesions between pre-discharge MR and follow-up MR (3 months later)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin - Cardiothoracic Department, Turin, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Barbero C, Ricci D, Cura Stura E, Pellegrini A, Marchetto G, ElQarra S, Boffini M, Passera R, Valentini MC, Rinaldi M. Magnetic resonance imaging for cerebral lesions during minimal invasive mitral valve surgery: study protocol for a randomized controlled trial. Trials. 2017 Feb 21;18(1):76. doi: 10.1186/s13063-017-1821-y. PMID 28222779